CLINICAL TRIAL: NCT02674100
Title: AHPBA Pancreatic Irreversible Electroporation (IRE) Registry for Pancreatic Cancer
Brief Title: American Hepato-Pancreato-Biliary Association (AHPBA) Pancreatic Irreversible Electroporation (IRE) Registry
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: The Americas Hepato-Pancreato-Biliary Association (Unknown)
Responsible Party: Principal Investigator, Robert C. Martin, Professor, University of Louisville
Other Study IDs: 06-326
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry

SUMMARY:
The purpose of this study is to create a registry to provide insight into treatment selection and treatment outcome of pancreatic IRE in order to develop an evidence base such that physicians can provide the best possible care to patients with pancreatic cancer requiring surgical interventions.

The investigators seek a better understanding of the uses of ablation in the treatment of unresectable soft tissue pancreatic tumors and the limitations, concerns and complications that earlier users have.

DETAILED DESCRIPTION:
Rationale:

The rationale for creating this multi-center clinical database is to optimally collect clinical and pathological data on patients with neoplasms in order to facilitate future clinical observational and outcomes-based research.

Inclusion Criteria

Patients will be considered eligible for inclusion into the database if they meet the following eligibility criteria:

Evidence/suspicion of Pancreatic neoplasm ≥ 18 years of age

Exclusion Criteria Patients will be considered ineligible for inclusion into the database if they are not able to give consent.

Inclusion of Women, Minorities and Vulnerable Subjects This protocol will include women and minority populations. Vulnerable subjects (prisoners, children, mentally disabled persons) will not be included in the study population.

Primary Study Objective(s):

To provide insight in treatment selection and treatment outcome of Pancreatic IRE in order to develop an evidence base such that physicians can provide the best possible care to patients with Pancreatic cancer requiring surgical intervention.

Secondary Study Objective(s):

To provide data on adverse events and complications related to IRE treatment.

The AHPBA will be responsible for data collection and will periodically audit the data for quality assurance purposes. The AHPBA will review outcomes reported by each participating Research Institution and if outcomes are in the lower percentile, the investigators will be offered support to analyze the reasons for the suboptimal outcomes and may seek support to improve outcomes. The participating Research Institutions will receive a certificate annually that acknowledges their participation in the Research Project.

Goal and Aims of Registry?

The Specific Aims are:

* Gain a better understanding of the uses of ablation in the treatment of unresectable soft tissue pancreatic tumors
* Understand the limitations, concerns, and complications that earlier users of ablation in the treatment of unresectable soft tissue pancreatic tumors have

Create a multi-institutional group that will both enroll in this registry study, but more importantly enroll in future, prospective ablation in the treatments of unresectable soft tissue pancreatic tumors studies. Any patient undergoing a soft tissue ablation may be included in this study. To confirm, you will always own your data and the registry will be used as data storage until you release your data for evaluation on a project-by-project basis.

What Patients are Eligible?

• Any patient to which the treating physician believes that ablation of their soft tissue would be feasible in the care of their disease.

Patients who can be followed and can provide outcome data to achieve the Goals and Aims of the Registry.

To participate, the only thing we need to obtain from your site is a regulatory approval letter stating that it is acceptable to collaborate with your patients de-identified data (sample data collection protocol is attached) and that you will be consenting your patients to this data collaboration (The Registry).

Case report forms/ data collection sheets are attached The data entry will be web based. All treatments must be entered-not just the first treatment. All follow up-up to 2 years or until death of patient-must be entered. Common follow up is every 3-4 months for first year and every 6 months for second year. In order to ensure data accuracy we require that, for the first 5 patients entered, the data sheets and their supporting documentation (de-identified labs, treatment dictation, etc.) be sent to us so we can make sure the data entry is correct and complete (e.g., lesion dimensions, measures of response or progression, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years of age) diagnosed with pancreatic cancer that are eligible for soft tissue ablation per the treating physician.

Exclusion Criteria:

* Have a cardiac pacemaker or ICD implant
* Non-removable implants with metal parts near target lesion
* Myocardial infarction within 3 months prior to enrollment
* Not suitable for general endotracheal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient greater than 18 years of age that the treating physician believes that ablation of their soft tissue would be feasible in the care of their pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 5 years
  Prospective collection of All Adverse Events that will be categorized as either IRE related or Non-IRE related and will be graded per CTCAE v4.0

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
  Capture overall survival in patients treated with IRE for their pancreatic tumors

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (16):
- United States (11):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - University of Colorado, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Atlantic Health, Millburn, New Jersey
  - Northwell Health Cancer Institute, Lake Success, New York
  - Gibbs Cancer Research, Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Methodist Digestive Institute, Dallas, Texas
- McGill University, Montreal, Quebec, Canada
- Sanno Hospital, Tokyo, Japan, Japan
- Centro Medico, Mexico City, Mexico
- National Taiwan University, Taipei, Taiwan
- Freeman Hospital, High Heaton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided